CLINICAL TRIAL: NCT03125018
Title: Accuracy of SpO2 for Noninvasive Pulse Oximeter Sensor (LNCS ADTX)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TR27479-TP16850A
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Results first posted 2017-07-28 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Test Subject (Experimental): All subjects are enrolled into the test group and receive the LNCS ADTX Sensor.
  Interventions: Device: LNCS ADTX Sensor

INTERVENTIONS:
Device: LNCS ADTX Sensor — Noninvasive pulse oximeter sensor.

SUMMARY:
In this study, the level of oxygen within the blood will be reduced in a controlled manner by reducing the concentration of oxygen the study volunteer breathes. The accuracy of a noninvasive pulse oximeter sensor will be assessed by comparison to the oxygen saturation measurements from a laboratory blood gas analyzer.

ELIGIBILITY:
Inclusion Criteria:

* Competent non-smoking adults between the ages of 18 and 40 for each series of tests.
* Subjects must understand and consent to be in the study.
* American Society of Anesthesiology Class 1 (Healthy subjects without any systemic disease at all).

Exclusion Criteria:

* Subjects who have any systemic disease at all.
* Subjects who do not understand the study and the risks.
* Smokers.
* Subjects who are pregnant.
* Subjects having either signs or history of peripheral ischemia.
* Others deemed ineligible by the clinical staff.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2014-09-30 (Actual); Primary Completion 2014-10-09 (Actual); Study Completion 2014-10-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test Subject
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Test Subject
Number analyzed (Participants) | 13
Age, Customized [Count of Participants; unit: Participants]
  20-37 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Sensor by Arms Calculation
Description: Accuracy will be determined by comparing the noninvasive blood oxygen saturation measurement of the pulse oximeter to that obtained from a blood sample and calculating the arithmetic root mean square error (Arms) value. In order to obtain the Arms value, the blood oxygen saturation measurement is subtracted from the pulse oximeter oxygen saturation measurement for a number of samples, the average of this difference is computed as the bias. The standard deviation of the differences is computed as the precision. The square root of the sum of the squares of bias and precision is computed as the Arms Error value.
Time Frame: 1-5 hours
Measure: Number; unit: % of oxygen saturated hemoglobin
Units Other Than Participants: data points
Arm/Group | Test Subject
Number analyzed (Participants) | 13
Number analyzed (data points) | 572
% of oxygen saturated hemoglobin | 2.0

ADVERSE EVENTS:
Arm/Group | Test Subject
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes